CLINICAL TRIAL: NCT04551274
Title: Investigating the Use of Virtual Music Therapy in Frontline Healthcare Workers During COVID-19
Brief Title: Music Therapy in Frontline Healthcare Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simon Fraser University (Other)
Collaborators: Music Heals Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Ryan D'Arcy, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H20-02015
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Mood; Emotional Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysts and Outcomes Assessors will be blinded to the group labels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Participants in the music therapy group will complete a 4 week music therapy program, with a minimum of 2 sessions per week.
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): Control group participants will not experience any intervention

INTERVENTIONS:
Behavioral: Music Therapy — Music Therapy interventions involve the use of live music (performed or created by the therapist and/or patient), and a process that includes patient-specific assessment, treatment, and evaluation
  Arms: Music Therapy

SUMMARY:
The objective of this project is to investigate the impacts of the COVID-19 pandemic on frontline healthcare workers, and determine if a virtual music therapy can improve mood and emotional state in this population.

For this pilot study, EEG will also be used to assess measures of functional connectivity, attention, and mood in adult participants. Participants will also be evaluated for measures of emotion using a standardized test battery (NIH toolbox).

This pilot study will show how frontline healthcare workers have been impacted by the COVID-19 pandemic, and provide evidence as to the effectiveness of Music Therapy to support mental health in this essential population.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to investigate (a) the self-described impact that the COVID-19 pandemic has had on frontline healthcare workers, and (b) the use of music therapy to improve mental healththis population. Built on top of our successful neuroscience and neuroimaging research, we aim to use behavioural assessments combined with portable EEG technology to monitor how metrics of brain function and mental health change over time in frontline healthcare workers undergoing Music Therapy.

Hypothesis:

We expect to see improvements in behavioural/emotional metrics as a result of music therapy - with correlations to changes in brain activation, markers of attention, and connectivity.

Justification:

Music Therapy interventions involve the use of live music (performed or created by the therapist and/or patient), and a process that includes patient-specific assessment, treatment, and evaluation. Music Therapy has shown to be effective in addressing symptoms related to global and social functioning in schizophrenia and/or serious mental disorders, gait and related activities in Parkinson's disease, depressive symptoms, and sleep quality.

Objectives:

1. The first objective of this study is to investigate how the COVID-19 pandemic has affected the lives of frontline healthcare workers
2. The second objective is to investigate the effect of music therapy on mental health in frontline healthcare workers during the COVID-19 pandemic
3. The third objective is to investigate EEG-related changes in frontline healthcare workers with music therapy, and correlate to behavioural changes

Research Design:

This is a longitudinal study design. 20 frontline healthcare workers will be recruited. 10 will be randomly assigned to no therapy (control) and 10 will be assigned to a music therapy (intervention) group. Random assignment will be prospectively performed using Microsoft Excel. Each subject code will be randomly assigned a decimal number from 0-1. All subject codes will then be sorted with their random numbers in ascending order. The 10 subject codes with the largest number will be placed in the intervention group, and the remaining 10 in the control group

Participants in the therapy group will complete 4 weeks of music therapy. Experimental measures will be completed before and after the 4 week period.

Statistical Analysis:

Outcomes from the EEG and behavioural assessments will be compared across groups and time points using a repeated Measures Analysis of Variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* All participants will be required to be frontline healthcare workers, (i.e. paramedics, EMTs, nurses, doctors). Participants will be adults aged 19 years and above, who are English speakers, with normal or corrected vision and hearing abilities. Participants will be required to have independent capacity to consent, as per Article 3.3 of the TCPS2. Due to the virtual nature of the study, participants will need to have access to a computer/laptop with a webcam to be able to interact with the music therapist and the study team.

Exclusion Criteria:

* Participants who have experienced a traumatic brain injury in the last 12 months, or who have previously been diagnosed with any other neurological, neuropsychological, or psychiatric diseases/disorders/conditions will not be enrolled in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in General Life Satisfaction score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Positive Affect score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Anger score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Fear score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Meaning & Purpose score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Sadness score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Emotional Support score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.
Change in Loneliness score - NIH Emotion Toolbox | 4 weeks
  The NIH Toolbox Emotion Battery is a comprehensive set of neuro-behavioral measurements that quickly assess emotional functions. It consists of surveys in the domains of Negative Effect ,Psychological Well-Being, Stress & Self-Efficacy, and Social Relationships. It is based on a nationally representative sample to enable cross-measure comparisons, and is well-suited for measuring outcomes in longitudinal studies. Questions for each subitem are arranged on a likert scale with associated scores from 1-5. The overall score for each measure (at each time point) is calculated as the sum of scores for each question.

SECONDARY OUTCOMES:
EEG - Change in power in the Delta band | 4 weeks
  Resting-state EEG will be recorded
EEG - Change in power in the Beta band | 4 weeks
  Resting-state EEG will be recorded
EEG - Change in power in the Alpha band | 4 weeks
  Resting-state EEG will be recorded
EEG - Change in power in the Theta band | 4 weeks
  Resting-state EEG will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Glen Chapman, PhD, Study Director — Simon Fraser University
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No